CLINICAL TRIAL: NCT05072886
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 1b Study Followed by an Open-Label Extension to Evaluate the Safety, Tolerability, and Preliminary Efficacy of Topical AT193 in the Treatment of Patients With Nail Psoriasis
Brief Title: Study of Efficacy and Safety of Investigational Treatment in Patients With Nail Psoriasis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azora Therapeutics Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Azora Therapeutics Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP01
Record Dates: First submitted 2021-09-29; First posted 2021-10-11 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Nail Psoriasis; Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AT193 (Experimental): Topical applied daily
  Interventions: Drug: AT193
- Placebo (Placebo Comparator): Topical applied daily
  Interventions: Drug: AT193

INTERVENTIONS:
Drug: AT193 — Topical applied to affected areas daily

SUMMARY:
Part 1 is a randomized, double-blind, placebo-controlled phase 1b study to evaluate AT193 in approximately 34 patients with nail psoriasis for 16 weeks. Part 2 is an open-label extension phase where all patients will receive active drug for an additional 16 weeks followed by a 2 week nontreatment period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nail psoriasis for at least 3 months preceding study entry
* Diagnosis or history of plaque psoriasis or psoriatic arthritis
* A female participant of childbearing potential must use appropriate contraceptive measures during the study period
* A female participant of childbearing potential must have a negative urine pregnancy test result at screening
* Written informed consent must be obtained before any study procedure is performed

Exclusion Criteria:

* Pregnant or breastfeeding
* Diagnosis of other active skin or nail diseases or skin or nail infections (bacterial, fungal, or viral) that may interfere with evaluation of skin or fingernail psoriasis
* History or evidence of a clinically significant disorder, condition, or disease that would pose a risk to patient safety or interfere with the study evaluation, procedures, or completion in the judgment of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sinclair Dermatology, East Melbourne, Victoria, Australia